CLINICAL TRIAL: NCT00992095
Title: A Single Dose, Two-Period, Two-Treatment, Two-Way Crossover Bioequivalency Study of Buprenorphine HCl (Sublingual) 8 mg Tablets With a Naltrexone Block Under Fasting Conditions
Brief Title: Bioequivalency Study of Buprenorphine Hydrochloride 8 mg Tablet Under Fasted Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Director - Drug Regulatory Affairs and Medical Affairs, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BUPR-T8-PVFS-1
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: buprenorphine hydrochloride — single dose 8 mg sublingual tablet
  Other Names: SUBUTEX

SUMMARY:
The objective of this study was to prove the bioequivalence of Buprenorphine HCl 8 mg tablet under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening.

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs. History of allergic or adverse response to buprenorphine hydrochloride or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2006-08; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
bioequivalence determined by statistical comparison Cmax | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Fredrick A. Bieberdorf, M.D., Principal Investigator — CEDRA Clinical Research
Locations (1):
- CEDRA Clinical Research, Austin, Texas, United States